CLINICAL TRIAL: NCT06582511
Title: Evaluating Metabolic Changes Induced by PhotoBioModulation (PBM) Through Spectrally Resolved Autofluorescence in Dry Age-Related Macular Degeneration (dAMD) Patients
Brief Title: Evaluating Metabolic Changes Induced by PhotoBioModulation Through Spectrally Resolved Autofluorescence in Dry Age-Related Macular Degeneration Patients
Acronym: PBM-dAMD
Status: Active, not recruiting | Type: Observational
Sponsor: Francesco Bandello (Other)
Responsible Party: Sponsor-Investigator, Francesco Bandello, Co-Investigator, IRCCS Ospedale San Raffaele
Organization: IRCCS Ospedale San Raffaele (Other)
Other Study IDs: PBM-dAMD
Record Dates: First submitted 2024-08-26; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Macular Degeneration, Age Related
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The best treatment to prevent the evolution of early and intermediate forms of dAMD to atrophic degeneration is PhotoBioModulation (PBM). It is based on the principle that molecules can absorb light even if it is not part of specialized light-receiving organs. Irradiation of cells at certain wavelengths can be used to activate native molecules to modulate biochemical reactions and, consequently, whole cellular metabolism. One of the main targets of PBM is mitochondrial activity. Mitochondria are sensitive to irradiation with red-NIR light. PBM might also function by increasing the bioavailability of nitric oxide (NO) by prompting its release from intracellular stores. It is proposed that PBM causes the photodissociation NO from CCO15. NO is known to inhibit electron transport, so dissociation of NO can increase the mitochondrial membrane potential, increase O2, consumption, and thus the proton gradient, ultimately leading to an increase in ATP production. NO can also diffuse outside and act as a messenger capable of causing vasodilation and other effects.

PBM demonstrated a beneficial role in dAMD, characterized by mitochondrial dysfunction, oxidative stress, and inflammation. SrAF allows to assess of mitochondrial function, a target of PBM, as it allows the observation of minor fluorophores such as FAD. The SrAF is used to evaluate the effectiveness of the treatment.

DETAILED DESCRIPTION:
This study is an observational, prospective, longitudinal, and monocentric study on Medical Device (CE marked, according to indications for use) on evaluating metabolic changes through Spectrally Resolved Autofluorescence in subjects with dry AMD.

Subjects will receive PBM treatments, as clinical practice, to stimulate metabolic mitochondrial activity which will be evaluated through Spectrally Resolved Autofluorescence.

Up to 30 subjects will be enrolled. The follow-up will last 6 months. Following the diagnosis of dAMD, the patient will be referred for photobiomodulation treatment.

Efficacy assessments will include slit lamp and fundus examinations, Intraocular pressure (IOP), ETDRS BCVA, CS, BAF, SR-AF, SD-OCT, Swept Source OCT-Angiography (SS-OCTA), and microperimetry. Whenever possible, the same person should perform the evaluations specified by the protocol at each study visit. Unless otherwise indicated, all ocular assessments should be performed on the study eye only.

Safety assessments include incidence of adverse events/serious adverse events, visual acuity, slit lamp findings, crystalline lens changes in phakic eyes, intraocular pressure, and fundus findings. The reporting period is from day 0 through the last study visit (Month 12).

The Primary Objective is to evaluate the modification of SrAF stimulated by the PBM treatment. The secondary objective is to evaluate the effectiveness of PBM treatment.

ELIGIBILITY:
INCLUSION CRITERIA

* Male or female at least 50 years;
* Subjects with ETDRS BCVA letter scores of between 50 and 80 (Snellen equivalent of 20/100 to 20/25);
* Subjects with a diagnosis of dry AMD as defined by the presence of drusen (regular or reticular pseudodrusen) and/or geographic atrophy (GA) visible on two of the following: color fundus images, OCT and/or Heidelberg FAF;
* Able to communicate well with the Investigator and able to understand and comply with the requirements of the study; The subject is informed of the nature of this study and has provided written informed consent in accordance with institutional, local, and national regulatory guidelines.

EXCLUSION CRITERIA

* Pregnant or lactating women
* Current or history of neovascular maculopathy that includes any of the following:

  * Macular neovascularization (MNV) is defined as pathologic angiogenesis originating from the choroidal vasculature that extends through a defect in Bruch's membrane
  * Serous and/or hemorrhagic detachment of the neurosensory retina or retinal pigment epithelial (RPE)
  * Retinal hard exudates
  * Subretinal and sub-RPE fibrovascular proliferation
  * Disciform scar
* Presence of center involving GA within the central ETDRS 500 μm diameter at diagnosis
* Media opacities, including cataracts, which might interfere with visual acuity or imaging in the study eye(s). Subjects should not be entered if there is likelihood that they will require cataract surgery in the study eye in the next 24 months
* Posterior capsule opacification, which might interfere with visual acuity or imaging in the study eye(s). Subjects should not be entered if there is likelihood that they will require surgery in the study eye in the next 24 months
* Invasive eye surgery (e.g. cataract, capsulotomy) on a qualifying eye within three 3 months before treatment
* Ocular disorder or disease that partially or completely obstructs the pupil (e.g., posterior synechia in uveitis)
* A visually significant disease in any ocular structure apart from dry AMD (e.g., diabetic macular edema, glaucoma (using >2 eye drops medications, uncontrolled IOP and/or central/paracentral visual field loss), glaucoma surgery, active uveitis, active vitreous disease, intraocular tumor, retinal vascular diseases)
* Has a serious medical illness that will prevent the subject from performing study activities (including cardiac, hepatic, renal, respiratory, endocrinologic, neurologic, or hematologic disease) or, in the judgment of the Investigator, is likely to require surgical intervention or hospitalization at any point during the study
* Presence of or history of malignancy within the past 5 years other than non-melanoma skin or squamous cell cancer or cervical carcinoma in situ
* Is non-ambulatory
* Presence or history of known light sensitivity to yellow light, red light, or near-infrared radiation (NIR), or if there is a history of light-activated CNS disorders (e.g., epilepsy, migraine)
* Use of any photosensitizing agent (e.g., topical, injectable) within 30 days of treatment without consulting the subject's physician
* History of drug, alcohol, or substance abuse within 3 months before treatment
* Has received an investigational drug or treatment with an investigational device within 3 months before treatment
* If on any antioxidant or vitamin Age-Related Eye Disease Study (AREDS) supplement for dry AMD, has not been stabilized for a minimum of 1 month before Screening. Subjects are considered to be stable if they are taking the AREDS supplements consistently as prescribed by their treating doctor.
* Has received Low Vision Rehab/Therapy within 30 days before Screening or intends to receive during the study
* In the opinion of the Investigator, is unlikely to comply with the study protocol

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 30 subjects will be enrolled from October 2021 to December 2023. The follow-up will last 6 months. Following the diagnosis of dAMD, the patient will be referred for photobiomodulation treatment. On the occasion of this visit, the patient will be offered to participate in the study.
  After providing informed consent and documenting it in writing, subjects will be screened.. Screening evaluations may be performed at any time within the 14 days preceding and subjects must fulfill the following criteria
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
changes in blue autofluorescence using Spectral Domain Optical Coherence Tomography (SD-OCT) | form baseline to month 6
  changes in blue autofluorescence using Spectral Domain Optical Coherence Tomography (SD-OCT
The change in SrAF To evaluate the modification of SrAF stimulated by the PBM treatment | from baseline until month 6
  evaluation of the changes in SrAF measurements

SECONDARY OUTCOMES:
Evaluation of changes in Best Corrected Visual Acuity (ETDRS) | form baseline to month 6
  Evaluation of changes in Best Corrected Visual Acuity (ETDRS)
Evaluation of changes in contrast sensitivity | form baseline to month 6
  Evaluation of changes in contrast sensitivity
evaluation of drusen volume, central drusen thickness, retinal volume, and central retinal thickness using Spectral Domain Optical Coherence Tomography (SD-OCT) | form baseline to month 6
  evaluation of drusen volume, central drusen thickness, retinal volume, and central retinal thickness using Spectral Domain Optical Coherence Tomography (SD-OCT)
evaluation of changes in choriocapillary perfusion density on Swept Source Optical Coherence Tomography Angiography (SS-OCTA) | form baseline to month 6
  evaluation of changes in choriocapillary perfusion density on Swept Source Optical Coherence Tomography Angiography (SS-OCTA)
evaluation of changes in retinal sensitivity on microperimetry and the rate of progression to advanced AMD (geographic atrophy) | form baseline to month 6
  evaluation of changes in retinal sensitivity on microperimetry and the rate of progression to advanced AMD (geographic atrophy)

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Ospedale San Raffaele, Milan, Italy/mi, Italy